CLINICAL TRIAL: NCT00659334
Title: Multi-disciplinary Study: MR, Histologic and EM Imaging of Intravenous Superparamagnetic Crystalline Particles (Combidex) to Brain, Intra-cerebral Tumors and in CNS Inflammation
Brief Title: Imaging of Intravenous (IV) Combidex to Brain, Intra-cerebral Tumors and in Central Nervous System (CNS) Inflammation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: AMAG not continuing with Combidex, the study drug
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Edward Neuwelt, Professor, OHSU Knight Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00001127; 5R01NS034608 (NIH); OHSU-1127 (Other: OHSU IRB)
Record Dates: First submitted 2008-04-10; First posted 2008-04-16 (Estimated); Results first posted 2012-11-09 (Estimated); Last update posted 2022-12-21 (Actual); Status verified 2022-11

CONDITIONS: Brain Neoplasms
Keywords: Combidex; Diagnostic imaging
MeSH Terms: conditions — Brain Neoplasms | interventions — ferumoxtran-10; Neurosurgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- 1 (Active Comparator): Adults with brain tumor to receive Combidex infusion only
  Interventions: Drug: Ferumoxtran-10 (Combidex)
- 2 (Active Comparator): Adults with brain tumors to receive Combidex infusion and neurosurgery
  Interventions: Drug: Ferumoxtran-10 (Combidex); Procedure: Neurosurgery
- 3 (Other): Adults with brain tumors to receive neurosurgery only (NO Combidex)
  Interventions: Procedure: Neurosurgery
- 4 (Active Comparator): Children with brain tumors to receive Combidex only
  Interventions: Drug: Ferumoxtran-10 (Combidex)
- 5 (Active Comparator): Children with brain tumors to receive Combidex and neurosurgery
  Interventions: Drug: Ferumoxtran-10 (Combidex); Procedure: Neurosurgery
- 6 (Other): Children with brain tumors to receive neurosurgery only, NO Combidex
  Interventions: Procedure: Neurosurgery
- 7 (Active Comparator): Adults with Inflammatory lesions (stroke or MS) to receive Combidex only
  Interventions: Drug: Ferumoxtran-10 (Combidex)

INTERVENTIONS:
Drug: Ferumoxtran-10 (Combidex) — 2.6 mg/kg
  Other Names: Combidex
  Arms: 1; 2; 4; 5; 7
Procedure: Neurosurgery — neuro-surgical tumor biopsy or resection to assess particle localization. Biopsy (stereotactic, when possible) will take place following the 24 hour post- Combidex MR and within 48 hrs of i.v. Combidex administration. Biopsies will be taken from the tumor, brain around tumor (BAT) and brain distant to tumor and the MR localization and histology will be compared. The tissue will be obtained by either resection or needle frameless stereotactic biopsy.
  Arms: 2; 3; 5; 6

SUMMARY:
Combidex (ferumoxtran-10) is an ultra-small iron oxide particle covered with a sugar coating. It has been evaluated as an MRI contrast agent for use in imaging well perfused organs such as the liver and spleen and for imaging lymph nodes. In this study, Combidex is being used to compare the standard imaging agent, Gadolinium, in imaging brain tumors and the area adjacent to the tumor location. Combidex may provide the ability to better see brain tumors and inflammatory lesions on magnetic resonance imaging (MRI) scans. Combidex may be useful in its ability to cross blood vessels into brain tumors, and because of its size and ability to get into the area next to brain tumors, could assist in the treatment of brain tumors with other drugs in the future.

DETAILED DESCRIPTION:
Subjects are recruited as patients in one of the neurology, neurosurgery or neuro-oncology clinics at OHSU. There are four groups of the study:

* Subjects receive the combidex infusion only.
* Subjects receive Combidex and undergo a previously schedule neurosurgery.
* Subjects undergo surgery only and provide a sample of their tumor tissue to be used in pathology studies of Combidex.
* Subjects with MS or stroke are invited to participate in receiving Combidex to evaluate the effectiveness of enhancing the area of damage within the brain.

Subjects are deemed eligible for the study and undergo a baseline MRI within 28 days of receiving Combidex. Subjects receiving Combidex are admitted for a half day into the Oregon Clinical & Translational Research Institute(OCTRI). Combidex is infused I.V. over 30 minutes. Subjects are monitored for side effects and are discharged within about 5 hours after the infusion, if no complications have been noted. Subjects return 24 hours after the infusion for a post infusion MRI scan and return again to one of the neurology clinics for one month follow-up. Subjects enrolled in group 2 undergo surgery 1-2 days after the Combidex infusion and also undergo a 24 post infusion MRI and return for one month follow-up. These subjects are also followed closely by the neurosurgical physician during the course of follow-up. Subjects enrolled in group 3 only undergo surgery and agree to have a piece of their tumor resection or biopsy donated for use in the study. Group 4 is the same as group 1, except the patient population includes multiple sclerosis and stroke instead of patients with brain tumors.

ELIGIBILITY:
Inclusion Criteria:

* Brain tumor or CNS inflammatory lesion including stroke or MS
* 5 yrs old or older
* Able to undergo MRI without general anesthesia
* Agree to be followed for 1 month following infusion of Combidex
* Sign a written informed consent
* If female and of child-bearing potential, be postmenopausal, sterile, or be on birth control for 1 month prior to study
* Must have a pre-treatment MRI within 28 days before study

Exclusion Criteria:

* Clinically significant signs of uncal herniation
* Allergy to study drug, Combidex
* Hepatic insufficiency
* Stage IV or V renal insufficiency
* If female, pregnant or lactating
* Require anesthesia for MRI scanning
* Hemachromatosis

Ages: 5 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2000-08; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward A Neuwelt, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects are recruited as patients in one of the neurology, neurosurgery or neuro-oncology clinics at OHSU.
Pre-assignment Details: There are seven groups in the study. In Groups 1(adults) and 4(pediatric) subjects receive the Combidex infusion only. In Groups 2(adult) and 5(pediatrics) subjects receive Combidex and undergo neurosurgery. In Groups 3(adult) and 6(pediatric) subjects undergo surgery with tissue exam; and in Group 7(adult only) subjects with MS or stroke.
Groups:
- Combidex Only (Group 1): Adults with brain tumor to receive Combidex infusion only
- Combidex and Neurosurgery (Group 2): Adults with brain tumors to receive Combidex infusion and neurosurgery
- Neurosurgery Only (Group 3): Adults with brain tumors to receive neurosurgery only (NO Combidex)
- Combidex Only (Group 4): Children with brain tumors to receive Combidex only
- Combidex and Neurosurgery (Group 5): Children with brain tumors to receive Combidex and neurosurgery
- Neurosurgery Only (Group 6): Children with brain tumors to receive neurosurgery only, NO Combidex
- Inflammatory Lesions (Group 7): Adults with Inflammatory lesions (stroke or MS) to receive Combidex only
Period: Overall Study
Arm/Group | Combidex Only (Group 1) | Combidex and Neurosurgery (Group 2) | Neurosurgery Only (Group 3) | Combidex Only (Group 4) | Combidex and Neurosurgery (Group 5) | Neurosurgery Only (Group 6) | Inflammatory Lesions (Group 7)
Started | 46 | 41 | 5 | 2 | 1 | 0 | 21
Completed | 38 (8 Screen failures) | 36 (5 Screen failures) | 5 | 2 | 1 | 0 | 20 (1 screen failure)
Not Completed | 8 | 5 | 0 | 0 | 0 | 0 | 1
Not completed — Screen Failure | 8 | 5 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: No eligible individuals were identified to enroll in Group 6.
Groups:
- Total: Total of all reporting groups
Arm/Group | Combidex Only (Group 1) | Combidex and Neurosurgery (Group 2) | Neurosurgery Only (Group 3) | Combidex Only (Group 4) | Combidex and Neurosurgery (Group 5) | Neurosurgery Only (Group 6) | Inflammatory Lesions (Group 7) | Total
Number analyzed (Participants) | 46 | 41 | 5 | 2 | 1 | 0 | 21 | 116
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 2 | 1 |  | 0 | 3
  Between 18 and 65 years | 37 | 35 | 5 | 0 | 0 |  | 19 | 96
  >=65 years | 9 | 6 | 0 | 0 | 0 |  | 2 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (13.2) | 48.4 (12.8) | 45.4 (14.2) | 14.7 (1.4) | 14.1 (0) |  | 43.0 (15.3) | 48.8 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 17 | 2 | 1 | 1 |  | 8 | 50
  Male | 25 | 24 | 3 | 1 | 0 |  | 13 | 66
Region of Enrollment [Number; unit: participants]
  United States | 46 | 41 | 5 | 2 | 1 |  | 21 | 116

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experience Optimal Imaging in Adult and Pediatric Brain Tumors to Establish Timing and Sequencing Parameters of Combidex.
Description: Signal intensity change in participants with Pre and 24 hours Post Combidex on T1, T2, T2* MRI sequences will be assessed (some patients undergo scans at 3 and 72 hours in order to assess radiographic changes at these time points). Combidex will be administered in dose 2.6 mg/kg in adults with high and low grade gliomas, metastases, meningiomas, and PNET; and in pediatric patients with astrocytomas grade i-iv, brain stem gliomas, ependymomas, CNS germ cell tumors, and PNET.
Time Frame: 24 hours (some patients between 3 and 72 hours) after administration of Combidex
Population: No eligible participants were identified to enroll in Group 6. Data not collected for Group 3 due to early study termination.
Measure: Number; unit: Participants
Arm/Group | Combidex Only (Group 1) | Combidex and Neurosurgery (Group 2) | Neurosurgery Only (Group 3) | Combidex Only (Group 4) | Combidex and Neurosurgery (Group 5) | Neurosurgery Only (Group 6) | Inflammatory Lesions (Group 7)
Number analyzed (Participants) | 46 | 41 | 0 | 2 | 1 | 0 | 21
Participants | 36 | 35 |  | 2 | 1 |  | 20

2. Secondary Outcome: Assess the Cellular Uptake of Particles in Brain Tumor Patients by Comparing Imaging Results With Histology and Electron Microscopic Examination of Biopsy Tissue
Time Frame: 2 years
Population: Data was not collected due to early study termination (Combidex became obsolete with introduction of ferumoxytol and this study was closed early).
Arm/Group | Combidex Only (Group 1) | Combidex and Neurosurgery (Group 2) | Neurosurgery Only (Group 3) | Combidex Only (Group 4) | Combidex and Neurosurgery (Group 5) | Neurosurgery Only (Group 6) | Inflammatory Lesions (Group 7)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Compare Combidex Imaging in Brain Tumor Patients, With Other CNS Inflammatory Lesions Such as Multiple Sclerosis and Stroke.
Time Frame: 2 years
Population: as for outcome 2
Arm/Group | Combidex Only (Group 1) | Combidex and Neurosurgery (Group 2) | Neurosurgery Only (Group 3) | Combidex Only (Group 4) | Combidex and Neurosurgery (Group 5) | Neurosurgery Only (Group 6) | Inflammatory Lesions (Group 7)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Compare Pre- and Post-op Gd Enhanced MRI Combidex Enhanced MR Imaging Done Pre-, Intra- and Post-operatively, to Assess the Degree of Resection and Residual Tumor.
Time Frame: 2 years
Population: as for outcome 2
Arm/Group | Combidex Only (Group 1) | Combidex and Neurosurgery (Group 2) | Neurosurgery Only (Group 3) | Combidex Only (Group 4) | Combidex and Neurosurgery (Group 5) | Neurosurgery Only (Group 6) | Inflammatory Lesions (Group 7)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: Other adverse events were collected/assessed, but none affected over 5% of the patient population.
Arm/Group | Combidex Only (Group 1) | Combidex and Neurosurgery (Group 2) | Neurosurgery Only (Group 3) | Combidex Only (Group 4) | Combidex and Neurosurgery (Group 5) | Neurosurgery Only (Group 6) | Inflammatory Lesions (Group 7)
Serious Adverse Events (participants affected / at risk) | 10/46 | 10/41 | 2/5 | 1/2 | 0/1 | 0/0 | 0/21
Other Adverse Events (participants affected / at risk) | 0/46 | 0/41 | 0/5 | 0/2 | 0/1 | 0/0 | 0/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combidex Only (Group 1) (N=46) | Combidex and Neurosurgery (Group 2) (N=41) | Neurosurgery Only (Group 3) (N=5) | Combidex Only (Group 4) (N=2) | Combidex and Neurosurgery (Group 5) (N=1) | Neurosurgery Only (Group 6) (N=0) | Inflammatory Lesions (Group 7) (N=21)
Disease Progression (Nervous system disorders) | 9 | 10 | 2 | 0 | 0 | 0 (0) | 0
Cerebellar Infraction (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 (0) | 0 — Cerebellar infraction in the left hemisphere.
Post-Op Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 (0) | 0 — Post-Op infection from craniotomy.

LIMITATIONS AND CAVEATS:
Early trial termination due to study drug Combidex no longer manufactured.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No